CLINICAL TRIAL: NCT07182292
Title: Effectiveness of Combined Therapeutic Exercise and Anti-Inflammatory Nutritional Supplementation in Frail, Malnourished Older Adults
Brief Title: Effect of a Combined Exercise and Anti-Inflammatory Nutritional Intervention in Frail Older Adults
Acronym: AliFrail
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Adventia Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AliFrail-HUN-2025
Record Dates: First submitted 2025-09-04; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Frail Elderly Syndrome; Malnutrition Elderly
Keywords: inflammaging; malnutrition; frailty
MeSH Terms: conditions — Malnutrition; Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Experimental - Combined Exercise + Anti-Inflammatory Supplement (Alisenoc™) (Experimental): Participants included in this group will perform physical exercise (Vivifrail) + Anti-Inflammatory Supplement
  Interventions: Dietary Supplement: Anti-Inflammatory Supplement
- Arm 2: Active Comparator - Exercise + Conventional Nutritional Supplement (Active Comparator): Participants included in this group will perform physical exercise (Vivifrail) + Conventional Nutritional Supplement
  Interventions: Dietary Supplement: Conventional Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: Anti-Inflammatory Supplement — A daily oral dose of Alisenoc™, an anti-inflammatory nutritional supplement specifically designed for older adults. Alisenoc™ contains olive oil polyphenols, omega-3 fatty acids (EPA/DHA), leucine-enriched protein, and antioxidant micronutrients to target inflammaging, sarcopenia, and nutritional deficiencies.
  Participants will be followed at 12 weeks, and at 6 and 12 months for functional, biochemical, and clinical outcomes.
  Arms: Arm 1: Experimental - Combined Exercise + Anti-Inflammatory Supplement (Alisenoc™)
Dietary Supplement: Conventional Nutritional Supplement — they will receive a conventional oral nutritional supplement that is isocaloric and protein-equivalent to the experimental product, but without anti-inflammatory ingredients.
  This standard supplement reflects routine nutritional support typically provided in geriatric clinical practice for malnourished patients. It contains energy, protein, and micronutrients but no specific anti-inflammatory components such as olive polyphenols or omega-3 fatty acids.
  Arms: Arm 2: Active Comparator - Exercise + Conventional Nutritional Supplement

SUMMARY:
The goal of this clinical trial is to evaluate whether a combined intervention of therapeutic exercise and anti-inflammatory nutritional supplementation improves physical performance and reduces systemic inflammation in frail, malnourished older adults. The main questions it aims to answer are:

Does the addition of an anti-inflammatory nutritional supplement (Alisenoc™) to a multicomponent exercise program (Vivifrail) lead to greater improvements in physical performance compared to standard exercise and conventional nutritional support?

Does the combined intervention reduce levels of inflammatory biomarkers (e.g., IL-6, TNF-α, IL-8, GDF-15) in this population?

Are there measurable changes in body composition (e.g., muscle mass, fat mass, bone health) following the intervention?

Does the intervention impact clinical outcomes such as hospital readmissions, functional independence, or mortality over the following 12 months?

Researchers will compare two groups:

One group receiving the Vivifrail exercise program plus a daily dose of the anti-inflammatory nutritional supplement Alisenoc™.

Another group receiving the same Vivifrail program plus an isocaloric, protein-equivalent conventional supplement.

Participants will:

Be aged 75 years or older and identified as frail and malnourished according to Fried and GLIM criteria.

Undergo baseline evaluation including functional performance (SPPB), body composition via bioimpedance analysis, and blood sample collection for inflammatory biomarkers.

Be randomly assigned to one of the two intervention groups.

Follow a 12-week home-based multicomponent exercise program guided by educational materials and supervised remotely.

Consume the assigned oral nutritional supplement daily for the same 12-week period.

Return for outcome assessments at 12 weeks, and again at 6 and 12 months for long-term follow-up.

All study procedures will take place at the Hospital Universitario de Navarra (HUN), Spain. Participants will be recruited from outpatient geriatrics and nutrition clinics and assessed at a dedicated research unit with nursing support. The intervention is designed to be feasible, scalable, and representative of real-world multidisciplinary care in older populations with high vulnerability.

The study aims to provide evidence for an integrative, personalized approach to reversing frailty through combined physical and nutritional strategies targeting the biological basis of inflammaging.

DETAILED DESCRIPTION:
Frailty and malnutrition are prevalent, closely interconnected syndromes in older adults, associated with adverse outcomes such as functional decline, falls, institutionalization, prolonged hospitalization, and increased mortality. These conditions reinforce each other in a bidirectional cycle: malnutrition contributes to muscle loss and diminished physical function, while frailty can lead to decreased appetite and nutrient intake. Both are increasingly linked to chronic, low-grade systemic inflammation, known as "inflammaging."

Inflammaging is characterized by persistently elevated levels of circulating pro-inflammatory cytokines, such as IL-6, TNF-α, IL-8, and CRP. This inflammatory environment contributes to sarcopenia, bone demineralization, insulin resistance, and immune system decline, all of which further drive the progression of frailty. Therefore, interventions that reduce inflammaging may offer a novel therapeutic pathway to mitigate frailty and its consequences.

Multicomponent physical exercise programs-especially those incorporating strength, balance, and endurance training-have demonstrated efficacy in improving mobility and reducing inflammation in older adults. The Vivifrail© program, developed and validated for frail and pre-frail populations, offers a structured, scalable home-based exercise model. At the same time, nutritional interventions enriched with anti-inflammatory ingredients-such as extra virgin olive oil polyphenols, omega-3 fatty acids (EPA/DHA), and leucine-may support muscle anabolism and reduce systemic inflammation. Yet, despite promising evidence from each modality alone, their combined impact in frail, malnourished populations remains understudied.

The AliFrail trial addresses this gap through a randomized, controlled, open-label, two-arm clinical study conducted at the Hospital Universitario de Navarra (HUN) in Pamplona, Spain. A total of 158 community-dwelling adults aged ≥75 years with frailty and malnutrition will be randomized to receive either:

1. the Vivifrail© exercise program plus a daily anti-inflammatory oral nutritional supplement (Alisenoc™), or
2. the same exercise program with an isocaloric, protein-equivalent standard nutritional supplement without anti-inflammatory components.

The intervention will last 12 weeks, followed by follow-up assessments at 6 and 12 months. The primary outcome is change in physical performance measured by the Short Physical Performance Battery (SPPB). Secondary outcomes include body composition (via bioelectrical impedance), inflammatory biomarker levels (IL-6, IL-8, TNF-α, GDF-15), handgrip strength, bone health (via REMS), quality of life (EQ-5D), and major clinical outcomes (readmissions, falls, mortality). Participant adherence, safety, and adverse events will also be monitored throughout the study period.

Sample size calculation is based on detecting a 1-point difference in SPPB between groups, assuming a standard deviation of 2 points, α = 0.05, and 80% power. This requires 158 participants in total, accounting for expected loss to follow-up.

Randomization will be stratified and computer-generated, with allocation concealed using sealed opaque envelopes. Due to the nature of the intervention, the trial will be open-label for participants and clinicians, but outcome assessors will remain blinded to minimize bias. Participants will be instructed not to reveal group allocation during assessments.

Data will be recorded in secure, encrypted electronic case report forms (eCRFs). Biological samples for biomarker analysis will be stored at -80°C. Data management procedures will ensure participant confidentiality and compliance with data protection regulations.

The study has been approved by the Research Ethics Committee of Navarra (CEIm Navarra). All participants (or legal representatives) will provide informed consent prior to enrollment. The trial will be registered on a public international platform (EU Clinical Trials Register) and conducted in accordance with SPIRIT 2013 guidelines, the Declaration of Helsinki, and Good Clinical Practice (GCP) standards.

Implementation Strategy:

While the Geriatrics and Nutrition departments at HUN are not formally integrated, they will jointly collaborate on patient recruitment and assessments, coordinated from a dedicated research consultation room with nursing support. This design allows implementation without disrupting existing clinical workflows.

Barriers to implementation include limited care pathway integration, participant mobility and cognitive challenges, and logistical complexities in supplement delivery. Facilitators include strong institutional support from HUN and Navarrabiomed, a multidisciplinary research team with prior experience in similar trials, and availability of infrastructure and staff for participant support.

Significance:

AliFrail is designed to generate high-quality evidence on a personalized, combined strategy to reverse frailty through physical and nutritional intervention. Its findings could influence future clinical guidelines and healthy aging policies by supporting scalable, multimodal approaches that address the underlying biology of frailty-namely inflammaging-while enhancing physical resilience and independence in vulnerable older adults.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 75 years.
* Diagnosis of frailty according to Linda Fried's criteria.
* Diagnosis of malnutrition according to GLIM (Global Leadership Initiative on Malnutrition) criteria.
* Barthel Index score ≥ 60 points.
* Absence of advanced chronic kidney disease (defined as glomerular filtration rate < 25 mL/min/1.73m²).
* Absence of terminal illness as defined by SECPAL (Spanish Society for Palliative Care) criteria.

Exclusion Criteria:

* Presence of type 1 or type 2 diabetes mellitus with poor metabolic control (HbA1c > 8% or insulin-dependent).
* Oropharyngeal dysphagia to liquids that prevents safe intake of oral supplementation.
* Moderate-to-severe cognitive impairment, defined as a score ≥ 5 on the Global Deterioration Scale (GDS) of Reisberg.
* Refusal to sign the informed consent by the patient, primary caregiver, or legal representative, or inability to obtain it.
* Known allergy or intolerance to any component of the study supplements.
* Institutionalized in a long-term care or residential facility.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | From baseline to 12 weeks after intervention start
  Change in physical performance assessed by the Short Physical Performance Battery (SPPB), a validated composite measure of lower extremity function. The SPPB includes three components: balance tests, gait speed, and repeated chair stands. Scores range from 0 to 12, with higher scores indicating better physical function and mobility.

SECONDARY OUTCOMES:
Phase Angle (PhA) | Baseline, 12 weeks
  Change in phase angle (degrees), calculated via vectorial bioimpedance analysis. (BIA 101 BIVA PRO, Akern Bioresearch, Italy).
Skeletal Muscle Mass Index (SMMI) | Baseline, 12 weeks
  Change in skeletal muscle mass index (kg/m²), calculated by dividing appendicular muscle mass (kg) by height squared (m²)
Inflammatory Biomarkers | Baseline and 12 weeks post-intervention
  Change in serum IL-6 concentration (pg/mL), IL-8 concentration (pg/mL), TNF-α concentration (pg/mL), and GDF-15 concentration (pg/mL) measured using immunoassay techniques (Olink)
Handgrip Strength (Jamar® Dynamometer) | Baseline, 12 weeks, post-intervention
  Change in upper body strength measured by maximum handgrip strength (kg) using a calibrated Jamar® dynamometer. Participants will perform three trials with their dominant hand, and the highest value in kilograms will be recorded. Higher values indicate better muscle strength.
Barthel Index Score | Baseline, 12 weeks, and 12 months post-intervention
  Change in functional independence as assessed by the Barthel Index, which measures basic activities of daily living (ADL) including feeding, bathing, dressing, and mobility. Scores range from 0 to 100, with higher scores indicating greater independence.
Lawton & Brody Instrumental Activities of Daily Living (IADL) Scale Score | Baseline, 12 weeks, and 12 months post-intervention
  Change in instrumental functional capacity as measured by the Lawton & Brody IADL Scale. This scale evaluates complex daily tasks such as managing finances, cooking, and using transportation. Scores range from 0 to 8, with higher scores
Fried's Frailty Phenotype Score | Baseline and 12 weeks post-intervention
  Change in frailty status measured using Fried's Frailty Phenotype, which assesses five criteria: unintentional weight loss, self-reported exhaustion, weakness (grip strength), slow walking speed, and low physical activity. The total score ranges from 0 to 5, where:
  0 = Robust,
  1-2 = Pre-frail,
  3-5 = Frail. Higher scores indicate greater frailt
EuroQol 5-Dimension 3-Level Questionnaire (EQ-5D-3L) Score | Baseline, 12 weeks post-intervention
  Change in self-perceived health-related quality of life, measured using the EuroQol 5-Dimension 3-Level (EQ-5D-3L) questionnaire. This instrument includes five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each with three levels of severity. The responses are converted into a single utility index score ranging from -0.594 to 1, where 1 indicates full health, 0 indicates death, and negative values indicate states worse than death.
Adherence, Safety, and Tolerability of the Intervention | Baseline, 12 weeks post-intervention
  Composite outcome including:
  Adherence: Percentage of scheduled exercise sessions and supplement doses completed during the 12-week intervention.
  Safety: Total number of adverse events (AEs) reported during the study period.
  Tolerability: Number of participants reporting intolerance or side effects related to exercise or supplementation.
  Retention: Percentage of participants who completed the study protocol (inverse of dropout rate).
  Each component will be analyzed descriptively and used to assess feasibility of the combined intervention.
Clinical Adverse Events: Readmissions, Falls, and Mortality | 12 weeks, and 12 months post-intervention
  Composite outcome tracking the following clinical events over a 12-month follow-up period:
  All-cause hospital readmissions (any unplanned hospital admission)
  Falls (as self-reported during monthly follow-up or documented in clinical records)
  All-cause mortality
  Each component will be analyzed separately as part of the overall safety and effectiveness assessment of the intervention.

IPD SHARING:
Plan to Share IPD: No